CLINICAL TRIAL: NCT06184074
Title: Effect of Aromatase Inhibitors on Lower Extremity Quantitative Ultrasonographic Measurements and Static and Dynamic Balance Scores in Breast Cancer Patients Using Aromatase Inhibitors
Brief Title: Effect of Aromatase Inhibitors on Ultrasonographic Measurements and Static and Dynamic Balance Scores in Breast Cancer
Status: Completed | Type: Observational
Sponsor: Sultan Abdulhamid Han Training and Research Hospital, Istanbul, Turkey (Other)
Responsible Party: Sponsor
Other Study IDs: 23-17
Record Dates: First submitted 2023-11-21; First posted 2023-12-28 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer; Aromatase Inhibitors; Balanced
Keywords: Aromatase Inhibitors; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Breast Cancer Patients Using Aromatase Inhibitors Group: Breast cancer patients using aromatase inhibitors at least 1 year
- Breast Cancer Patients Group: Breast cancer patients who have not used aromatase inhibitors before

SUMMARY:
To evaluate the effects of aromatase inhibitors on lower extremity ultrasonographic measurements, static and dynamic balance scores in breast cancer patients using aromatase inhibitors

DETAILED DESCRIPTION:
Breast cancer is the most common cancer in women. 2/3 of breast cancer patients are estrogen and progesterone receptor positive. Tamoxifen or aromatase inhibitors are preferred in most of these patients depending on menopausal status. The increase in the life expectancy of breast cancer patients with medical treatments pushes us to find the cause of the drug side effects encountered during this extended life span and work on preventing/correcting them. It has been proven that aromatase inhibitors cause arthralgia in 40-50% of patients and a loss in bone mineral density, leading to a tendency towards osteoporosis. In this patient group, changes in the tendon and tendon sheath were also observed in ultrasonographic and magnetic resonance imaging and were stated to be the cause of the current symptoms.

In the literature, breast cancer patients have been evaluated in detail in terms of balance, and it has been shown that static and dynamic body balance is worse in this group compared to the control group. Among the breast cancer population, the presence of arthralgia in the patient group using aromatase inhibitors causes an increased risk of falls. In addition, it is thought that lower extremity tendon changes may be a factor in balance and proprioception disorders.

Based on this information, quantitative evaluation of static and dynamic balance in patients is important since there is an increase in the frequency of falls and a tendency to osteoporosis in patients using aromatase inhibitors in breast cancer. No similar study has been found in the literature.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal Woman
* Between 40-70 ages
* Stage 1-3 breast cancer
* Chemotherapy treatment due to breast cancer (Last dosage at least 6 months ago)
* Using an aromatase inhibitors for at least 1 year for group 1
* Never using an aromatase inhibitors at all for group 2
* Volunteers must sign and agree to participate in the study.

Exclusion Criteria:

* Stage 4 breast cancer
* Having active chemotherapy
* Older age patient (over 70 years old)
* Using of steroid
* Presence of diabetes mellitus that lasts longer than 3 years or insulin usage
* Neuropathic complaints
* Lack of vitamin B12 and thyroid dysfunction
* Dn4 (dolour neuropathic 4 question) score of 4 and above
* History of stroke
* Presence of polyneuropathy diagnosis
* Medication due to polyneuropathy diagnosis (gabapentin, pregabalin, duloxetine)
* Loss of motor function in the lower extremity
* Use of assistive devices for walking
* Presence of vestibular disorder
* Presence of cognitive impairment

Ages: 40 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Postmenopausal woman with breast cancer, between 40-70 years old
Sampling Method: Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Biodex Balance System | 5 months
  We will evaluate the patients with Limit of Stability test (LOS) protocols in the biodex balance system. For these tests, the rules specified in the Biodex guide will be applied and the results will be compared between two groups
Biodex Balance System | 20 weeks
  We will evaluate the patients with Fall Risk Test protocols in the biodex balance system. For these tests, the rules specified in the Biodex guide will be applied and the results will be compared between two groups
Biodex Balance System | 21 weeks
  We will evaluate the patients with Postural Stability Test protocols in the biodex balance system. Biodex guide will be applied and the results will be compared between two groups.

SECONDARY OUTCOMES:
Time Up and Go test (TUG) | 6 months
  Time Up and Go test (TUG) will be used to determine dynamic balance.A performance longer than 12 seconds indicates an increased risk of falling.
Brief Pain Inventory | 20 weeks
  . Brief Pain Inventory determines the severity of pain, each question is scored out of 10 and the average is calculated. A score of 10 is indicative of the worst pain
Tinetti Balance and Gait Test | 21 weeks
  It will be used to determine the risk of falling. The maximum score is 35. High values indicate good balance.
Fall Efficiency Scale | 22 weeks
  Fall Efficiency Scale will be used to evaluate the fear of falling, and this test is a scale that evaluates patients' fears of falling. It consists of 10 questions scored out of 10. A score above 70 indicates a high fear of falling.
Womac pain index (The Western Ontario and McMaster Universities Arthritis Index) | 20 weeks
  Womac index: It consists of 24 different questions in 3 different categories. Each answer is scored between 0-4. 4 indicates the worst pain state.
The European Organization for Research and Treatment of Cancer breast cancer module (EORTC QLQ-BR23) | 18 weeks
  It is a breast-specific module consisting of 23 questions to evaluate discomfort caused by breast cancer. Body image will be evaluated.
The European Organization for Research and Treatment of Cancer breast cancer module (EORTC QLQ-BR23) | 25 weeks
  It is a breast-specific module consisting of 23 questions to evaluate discomfort caused by breast cancer. Future perspective will be evaluated.
The European Organization for Research and Treatment of Cancer breast cancer module (EORTC QLQ-BR23) | 24 weeks
  It is a breast-specific module consisting of 23 questions to evaluate discomfort caused by breast cancer. Breast symtoms will be evaluated.
The European Organization for Research and Treatment of Cancer breast cancer module (EORTC QLQ-BR23) | 22 weeks
  It is a breast-specific module consisting of 23 questions to evaluate discomfort caused by breast cancer. Arm symtoms will be evaluated.
The European Organization for Research and Treatment of Cancer Core module EORTC-QLQ-C30 | 23 weeks
  It is a module consisting of 30 questions to evaluate discomfort caused cancer.
The European Organization for Research and Treatment of Cancer breast cancer module (EORTC QLQ-BR23) | 6 months
  It is a scale designed to evaluate functional status in breast cancer patients.
Patellar Tendon Ultrasound | 23 weeks
  The short axis of the ultrasound probe will be placed in the vertical plane, 6 mm below the lower pole of the patella and the patellar tendon will be imaged with ultrasound. Echogenicity will be calculated by uploading the image to the image j system. Lower values of echogenicity will indicate worse tendon quality
Patellar Tendon Ultrasound | 22 weeks
  The patellar tendon will be visualized by placing its long axis in a vertical plane 6 mm below the lower pole of the patella. Tendon thickness will be measured from this location(mm)
Quadriceps Tendon Ultrasound | 20 weeks
  The short long of the ultrasound probe will be placed in the vertical plane, 10 mm above the upper pole of the patella.Tendon thickness will be measured from this location(mm)
Quadriceps Tendon Ultrasound | 22 weeks
  The short axis of the ultrasound probe will be placed in the vertical plane, 10 mm above the upper pole of the patella.Echogenicity will be calculated by uploading the image to the image j system.Lower values of echogenicity will indicate worse tendon quality
Achilles tendon ultrasound | 21 weeks
  The short axis of the ultrasound probe will be placed in a vertical plane 2 cm above the distal calcaneus and the Achilles tendon will be visualized with ultrasound.Echogenicity will be calculated by uploading the image to the image j system.Lower values of echogenicity will indicate worse tendon quality.
Achilles tendon ultrasound | 20 weeks
  The short axis of the ultrasound probe will be placed in a vertical plane 2 cm above the distal calcaneus and the Achilles tendon will be visualized with ultrasound.Tendon thickness will be measured from this location(mm)

CONTACTS AND LOCATIONS:
Overall Officials: Ece Küçük, Principal Investigator — Sultan 2. Abdulhamid Han Training and Research Hospital
Locations (1):
- Ece Küçük, Istanbul, Turkey (Türkiye)